CLINICAL TRIAL: NCT04198233
Title: Impact of Placement of a Diazepam Suppository Intraoperatively on Early Postoperative Pain Following Pelvic Reconstructive Surgery: a Double-Blind, Randomized Placebo-Controlled Trial
Brief Title: Impact of Placement of a Diazepam Suppository on Early Postoperative Pain Following Pelvic Reconstructive Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 19-130
Record Dates: First submitted 2019-12-11; First posted 2019-12-13 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2019-12

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Diazepam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: All surgeons, patients and research staff will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Diazepam group (Experimental): Rectal Diazepam suppository
  Interventions: Drug: Diazepam
- Placebo group (Placebo Comparator): Placebo suppository
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Diazepam — Diazepam 10 mg compounded suppository
  Arms: Diazepam group
Drug: Placebos — Placebo suppository
  Arms: Placebo group

SUMMARY:
This is a randomized double-blinded placebo controlled trial to examine the use of rectal diazepam suppositories after major vaginal pelvic organ prolapse surgery will decrease postoperative pain in the interval between 3.5 and 6 hours postoperative compared to placebo.

DETAILED DESCRIPTION:
Hysterectomy is the most common major surgery performed in gynecology. Minimally invasive techniques for hysterectomy including vaginal and laparoscopic routes are preferred over the more invasive abdominal procedures, which are associated with more pain, longer hospital stays, and increased rates of complications.

Research has continued to provide evidence that same day discharge (SDD) after hysterectomy is safe, cost effective, and well received by patients. Pain is a common concern for patients undergoing major pelvic surgery and pain must be well controlled prior to discharge home.

Rectal administrations of medications are an attractive option postoperatively in patients desiring SDD. Rectal analgesia avoids 1st pass metabolism in the liver, leading to increased bioavailability of many medications and fewer side effects such as nausea and vomiting.

The purpose of the study is to investigate whether perioperative administration of a rectally administered diazepam suppository results in improved pain scores between 3.5 and 6 hours postoperatively in patients undergoing major vaginal pelvic reconstructive surgery.

ELIGIBILITY:
Inclusion Criteria:

* English speaking, able to understand informed consent and questionnaires
* Vaginal hysterectomy with vaginal vault suspension by one of the providers in the Division of Urogynecology and Reconstructive Pelvic Surgery at TriHealth, Inc.

  * With or without anterior and posterior repairs
  * With or without concomitant procedure for stress urinary incontinence
  * With or without removal of fallopian tubes or ovaries

Exclusion Criteria:

* Use of mesh for prolapse repair
* Robotic, laparoscopic, or open technique used for prolapse repair and/or hysterectomy
* Concomitant procedure done by an additional surgeon
* Concomitant anal sphincteroplasty or rectovaginal fistula repair
* Contraindication to use of Diazepam:

  * Allergy to Diazepam or other benzodiazepines
  * Acute narrow-angle glaucoma
  * Untreated open-angle glaucoma
  * Myasthenia gravis
  * Severe respiratory impairment
  * Severe hepatic impairment
* History of chronic pelvic pain receiving medical care
* Daily use of medication for pain: NSAID, Tylenol, opioid, gabapentin, and/or amitriptyline
* Pregnancy

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2020-02-12 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Vaginal/Rectal pain in Visual Analogue Scale (VAS) score | between 3.5 and 6 hours postoperatively
  VAS is a validated 100 millimeter scale with no pain as 0 mm and worst pain as 100 mm. Subjects draw a vertical line on the scale corresponding to their pain level.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Pauls, MD, Principal Investigator — TriHealth - Cincinnati Urogynecology Associates
Locations (1):
- Trihealth (Good Samaritan Hospital, Bethesda North Hospital), Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Aldrich ER, Tam TY, Saylor LM, Crisp CC, Yeung J, Pauls RN. Intrarectal diazepam following pelvic reconstructive surgery: a double-blind, randomized placebo-controlled trial. Am J Obstet Gynecol. 2022 Aug;227(2):302.e1-302.e9. doi: 10.1016/j.ajog.2022.05.009. Epub 2022 May 10. PMID 35550374